CLINICAL TRIAL: NCT03040544
Title: Efficacy of Goal-directed Minimally Invasive Surgery Simulation Training With the Lübeck Toolbox-Curriculum Prior to First Operations on Patients: Study Protocol for a Multi-centre Randomized Controlled Validation Trial (NOVICE)
Brief Title: Goal-directed MIS Simulation Training With the LTB-Curriculum Prior to First Operations on Patients: Study Protocol for a Multi-centre Randomized Controlled Validation Trial (NOVICE)
Acronym: NOVICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Michael Thomschewski, Dr., University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NOVICE trial
Record Dates: First submitted 2017-01-29; First posted 2017-02-02 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Minimally Invasive Surgery Basic Skills
Keywords: minimally invasive surgery; video-based trainer; laparoscopic; simulation training; surgical education
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTB-Curriculum (Experimental): First group/arm undergo MIS training according to the LTB curriculum after the first own laparoscopic cholecystectomy in the OR as a baseline. After 6 weeks, the participants in this group/arm will perform their second CHE. The video recordings of the MIS procedures will be analysed and compared using the Global Operational Assessment of Laparoscopic Skill (GOALS) score.
  Interventions: Procedure: LTB-Curriculum; Procedure: Laparoscopic cholecystectomy
- no LTB-Curriculums (Active Comparator): Second group/arm will not undergo any MIS trains after their first laparoscopic CHE in the OR. After 6 weeks, the participants in this group/arm will perform their second CHE. The video recordings of the MIS procedures will be analysed and compared using GOALS score.
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: LTB-Curriculum — The Lübeck Toolbox (LTB) curriculum has a structured training program, in which the laparoscopic basic skills are to be learned in six consecutive exercises. In doing so, the curriculum has precise targets for each of the six exercises based on the abilities of 15 MIS experts as a benchmark. The LTB curriculum is thus a structured training program with clear objectives that enable the technical learning of MIS basic skills comparable to the expert level.
  Arms: LTB-Curriculum
Procedure: Laparoscopic cholecystectomy — Performing Laparoscopic cholecystectomy by surgical residents without previous experience in MIS

SUMMARY:
Background: Laparoscopic surgical procedures have become increasingly established in operative medicine. They require special motor, haptic, and spatial-visual skills to perform the interventions safely and effectively. These minimally invasive surgery (MIS) basic skills are often learned in the operating room (OR) on the patient. This is economically inefficient and can be improved with regard to patient safety. Against the background of this problem, various simulators and video-box trainer have been developed in order to train laparoscopic basic skills outside the OR. The Lübecker Toolbox (LTB) curriculum is a video-based trainer including standardized and validated exercises with defined targets, based on the skills of experts MIS. Conducting MIS training outside the OR prior to performing the first MIS procedures on patients could be a sensible and valuable contribution to effective surgical education. An evidence of effectiveness in the practice transfer could have a considerable relevance with regard to the integration of MIS training programs into surgical education programs.

Aim of the study: The aim of the study is to investigate whether surgical residents without previous active experience in MIS are able to improve laparoscopic skills in MIS procedures in the OR, if they have successfully completed the LTB curriculum.

In the multicentric prospective study, will be conducted with surgical residents (SR) without prior active experience in MIS (n=14). After the SR have completed their first laparoscopic cholecystectomy (CHE), they will be randomized into two groups: 1) The intervention group will perform the LTB-Curriculum, whereas 2) the control group will not undergo any MIS training. After 6 weeks, both groups will perform the second laparoscopic CHE. Improvements in operative performance (between CHE I and CHE II) will be evaluated according to the Global Operative Assessment of Laparoscopic Skill (GOALS) Score (primary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* no motor or sensory restrictions when using surgical instruments surgical instruments.
* no previous performed MIS simulation training
* no previous performed MIS procedure ( any previous assisted MIS procedures are not an exclusion criterion)
* residents in surgical education for general or visceral surgery in Germany

Exclusion Criteria:

* The participant are not allowed to perform any other MIS training programs during the study period
* Before the start of the study, participants are not allowed to have performed any prior MIS simulation training or any MIS procedure

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-05-22 (Actual); Primary Completion 2020-05-21 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Global Operative Assessment of Laparoscopic Skill (GOALS)-Score | end of inclusion of all participants
  The GOALS score is an internationally established score for evaluating the MIS skills of a surgeon

SECONDARY OUTCOMES:
operation time | 8-12 weeks
  operation time of CHE I and CHE 2
percentage of the participants operating time in the total time of the CHE | 8-12 weeks
  percentage of participants operating time in the total time of the CHE I and CHE II
number of takeovers by the specialist assisting the CHE | 8-12 weeks
  experienced consultant surgeon will assist the CHE. The specialist can take over the operation at any time and perform surgical steps independently, according to his/her judgement with regard to the individual situation
potential conversion to laparotomy | 8-12 weeks
  potential conversion of the MIS CHE to open surgery

OTHER OUTCOMES:
sex of participant | 8-12 weeks
  sex of participant (male or female)
dominant hand of participant | 8-12 weeks
  dominant hand of participant (right or left)
age of participant | 8-12 weeks
  age of the participants
correlation with activities and hobbies | 8-12 weeks
  in particular playing an instrument, handicrafts and computer games
inter-rater reliability | 8-12 weeks
  possible differences and bias between video ratings by calculation

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Benecke, MD, Study Director — Medical University Center Schleswig-Holstein Campus Lübeck; Tilman Laubert, MD, Study Director — Medical University Center Schleswig-Holstein Campus Lübeck
Locations (1):
- Medical University Center Schleswig-Holstein Campus Lübeck, Department of surgery, Lübeck, Schleswig-Holstein, Germany